CLINICAL TRIAL: NCT00205491
Title: Pharmacological Intervention in Depression After Traumatic Brain Injury (A Research Study Within the Traumatic Brain Injury Model System)
Brief Title: Pharmacological Intervention in Depression After Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H133A02051602; H133A020516
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: depression after brain injury; traumatic brain injury; Venlafaxine
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: Venlafaxine

SUMMARY:
The purpose of this study is to determine if treatment with venlafaxine reduces symptoms of depression in persons with traumatic brain injury.

DETAILED DESCRIPTION:
The study evaluates the benefits of a promising antidepressant medication for the treatment of persons with traumatic brain injury (TBI) and major depressive disorder (MDD). The study is a randomized, double-blind, placebo-controlled trial of venlafaxine (a serotonin and norepinephrine reuptake inhibitor, also known as Effexor). Venlafaxine has been well established in the treatment of MDD in healthy individuals and is a recommended depression treatment agent for persons with TBI. By using a rigorous scientific methodology, this study will be an important first step in advancing the treatment of depression in this population beyond general impressions to proven treatments.

ELIGIBILITY:
Inclusion Criteria:

* Must have a documented traumatic brain injury (TBI), defined as damage to brain tissue caused by an external mechanical force as evidenced by: loss of consciousness due to brain trauma, or post traumatic amnesia (PTA), or skull fracture, or objective neurological findings that can be reasonably attributed to TBI on physical examination or mental status examination.
* Age 18 years or older
* At least three months postinjury
* Presence of major depressive disorder (MDD), as defined by Structured Clinical Interview for DSM-IV (SCID) interview
* Hamilton Depression Rating Scale (Ham-D) scores of 18 or greater on two consecutive evaluations (screening and baseline)

Exclusion Criteria:

* Individuals under 18 years of age
* Pregnancy, as determined by urine pregnancy screen
* Prisoners
* Individuals who are institutionalized
* Individuals who are not cognitively capable of completing the SCID interview and the Ham-D
* Unstable medical condition, defined as any significant medical condition likely to require hospitalization during the study period, or requiring adjustment in medications in the past month
* Active suicidality
* Severe depression that, in the investigator's professional opinion, will likely require hospitalization during the study time period
* Diagnosis of bipolar disorder, as defined by SCID interview
* Diagnosis of schizophrenia or other psychotic disorder, as defined by SCID interview, other than major depression with psychotic features
* Active drug or alcohol abuse within the past 3 months, as defined by SCID interview
* Dysphagia sufficient to preclude use of oral medications
* Known hypersensitivity to venlafaxine
* Use of monamine oxidase inhibitors (MAOI) within the past month
* Treatment with antidepressant medication within the past 3 months
* Concomitant administration of medications that interact with venlafaxine to a clinically significant degree

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Score on the Hamilton Rating Scale for Depression (Ham-D)at 12 weeks.

SECONDARY OUTCOMES:
Scores on cognitive and psychomotor tests at 12 weeks.
Scores on a satisfaction with life measure and a functional measure at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Kreutzer, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States